CLINICAL TRIAL: NCT00223756
Title: VA Low Vision Intervention Trial
Acronym: LOVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C3457-R
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Vision, Low
Keywords: Vision, Low
MeSH Terms: conditions — Vision, Low | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): interdisciplinary, outpatient blind rehabilitation
  Interventions: Other: Low Vision Intervention - Outpatient Training Program
- Arm 2 (No Intervention): usual care

INTERVENTIONS:
Other: Low Vision Intervention - Outpatient Training Program — Patients receive LV therapy as outpatients
  Other Names: Therapy Group
  Arms: Arm 1

SUMMARY:
The primary purpose of this research study is to evaluate the effectiveness of a new outpatient low vision rehabilitation program that is targeted to serve legally blind veterans with central vision loss. The hypothesis is that veterans in the treatment group will self-report less difficulty performing daily activities than veterans in the control group who are on a waiting list for VA low vision or blind rehabilitation programs.

DETAILED DESCRIPTION:
Abstract: Research Question:

Estimates are that there will be 854,000 severely visually impaired veterans in the year 2005 and 890,000 in the year 2010. Statistics, based upon the 2000 census, suggest that it will be well into the next decade before the number of severely visually impaired veterans begins to decrease. Waiting time for admission to VA blind rehabilitation centers (BRCs) is often a year or more. Low vision services are an important aspect of blind rehabilitation, as 85% of veterans admitted to BRCs have useful remaining vision. In the private sector, low vision services are provided in outpatient settings. Yet, legally blind veterans are still encouraged, if not required, to attend regional inpatient programs to obtain therapy with low vision devices because a reimbursement model is not available for outpatient blind rehabilitation and few low vision outpatient clinics have rehabilitation professionals to provide this training. The VA system needs alternative service delivery options for veterans who are unable to participate in inpatient rehabilitation. Outpatient low vision programs should provide continuity of care with the regional BRC programs and insure local access to low vision care that is high quality, timely, and cost-effective. Currently, the VERA Reimbursement Model allocates $27,826 per blind rehabilitation admission. Outpatient low vision programs have the potential to substitute for inpatient low vision services and more costly inpatient rehabilitation programs may not be necessary for higher functioning veterans. The purpose of the proposed research is to measure the effectiveness of a low vision outpatient program for legally blind veterans with central vision loss from macular diseases that could be provided at local VA facilities.

Specific Objectives are to:

1. Compare the mean change in self-report of difficulty performing daily activities measured with the Veteran's Affairs Low Vision Visual Function Questionnaire - 48 (VA LV VFQ-48) reading domain scores from baseline to 4 months after randomization [two months after veterans participate in a low vision outpatient program or usual care (waiting list) control group].
2. Determine if the mean change in VA LV VFQ-48 composite and reading domain scores from baseline to 4 months after randomization [two months after veterans participate in a low vision outpatient program or usual care (waiting list) control group] can be predicted by baseline measures of visual impairment, functional status and life state or explained by measures of functional status after rehabilitation.
3. Perform an economic evaluation of costs and cost-effectiveness of the low vision outpatient program.
4. Compare the mean change in VA LV VFQ-48 scores from the clinical trial from baseline to 4 months after randomization (two months after veterans participate in a low vision outpatient program) to historical data on the mean change in VA LV VFQ-48 scores from the Hines BRC program.

Hypothesis: Compared to the usual care (waiting list) control group, veterans in the treatment group will self-report a reduction of .78 logits or more in difficulty performing daily living activities measured by the VA LV VFQ-48 reading domain scores from baseline to 4 months after randomization (two months after veterans participate in a low vision outpatient program).The .78 logit change is clinically significant, as this improvement corresponds to the change in visual ability that would accompany a 6-line improvement on an EDTRS visual acuity chart.

Significance: The NIH includes visual impairment, chronic visual deficiencies that impair everyday function that are not correctable by ordinary glasses, among the 10 most prevalent causes of disability in America. Persons confronted with vision loss often feel limited and frustrated performing everyday activities such as reading, traveling from place to place, and recognizing objects or people. As a result, they may experience loss of self esteem, social isolation, difficulty working and reduced independence. The low vision team evaluates the level of remaining vision, prescribes special lenses or devices and techniques for using remaining vision more effectively. Low vision rehabilitation restores independence by enabling persons with vision loss to perform daily living tasks independently at home, at work or within the community.

Research Design: the proposed study is a randomized clinical trial conducted at two sites. Subjects are 122 legally blind veterans from Hines Hospital and Heffner VAMC. Veterans will be randomized to treatment from a new low vision outpatient program or a usual care (waiting list) control group. Following a low vision examination, veterans in the treatment group will receive 5 (2-2 1/2 hour) therapy sessions at the local VA sites and one home visit to evaluate the home environment and set up prescribed devices. The primary outcome measure is change in reading domain scores on the VA LV VFQ-48, a telephone questionnaire where subjects self-report their difficulty performing daily living activities in the community. Other measures include, instructors rating of veteran's visual skills and use of low vision devices after rehabilitation, visual skills for reading (PEPPER VSRT), health status (SF-36), and symptoms of depression (CES-D). Outcomes will be compared with T tests. Multiple linear regression models will be used to identify predictors and explain outcomes. Costs and cost effectiveness of outpatient treatment compared to treatment in an inpatient BRC will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Primary eye diagnosis (in better seeing eye) of either macular degeneration, macular dystrophy, macular hole or inflammatory disease of the macula
2. Habitual visual acuity (in better seeing eye) better than 20/500 but less than 20/100

Exclusion Criteria:

1. does not have a phone
2. does not speak English
3. has previously received low vision services as part of an inpatient blind rehabilitation program
4. has participated in a low vision program that provided low vision devices to meet reading needs with low vision therapy administered by an occupational therapist or vision rehabilitation professional since most recent significant decrease in vision
5. has English literacy less than 5th grade level
6. has habitual visual acuity in better seeing eye of equal to or better than 20/100, less than or equal to 20/500
7. fails Telephone Interview of Cognitive Status (TICS) screening (score of 30 or lower)
8. has history of stroke with aphasia
9. has other health condition that would preclude follow-up (e.g. significant malignancy or life-threatening disease)
10. is unable or unwilling to attend clinic visits required for the study
11. has severe hearing impairment that interferes with participation in telephone questionnaires
12. reports significant loss of vision since last eye exam
13. has vitreous hemorrhage, serous or hemorrhagic detachment of the macula, clinically significant macular edema or cystoid macular edema that is likely to result in further loss or improvement in vision after treatment in better seeing eye
14. plans cataract extraction in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
VA LV VFQ-48 Reading Domain Scores | 4 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joan Stelmack, OD MPH, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Result] Stroupe KT, Stelmack JA, Tang XC, Reda DJ, Moran D, Rinne S, Mancil R, Wei Y, Cummings R, Mancil G, Ellis N, Massof RW. Economic evaluation of blind rehabilitation for veterans with macular diseases in the Department of Veterans Affairs. Ophthalmic Epidemiol. 2008 Mar-Apr;15(2):84-91. doi: 10.1080/09286580802027836. PMID 18432491
- [Result] Stelmack JA, Tang XC, Reda DJ, Rinne S, Mancil RM, Massof RW; LOVIT Study Group. Outcomes of the Veterans Affairs Low Vision Intervention Trial (LOVIT). Arch Ophthalmol. 2008 May;126(5):608-17. doi: 10.1001/archopht.126.5.608. PMID 18474769
- [Result] Stelmack JA, Tang XC, Reda DJ, Moran D, Rinne S, Mancil RM, Cummings R, Mancil G, Stroupe K, Ellis N, Massof RW. The Veterans Affairs Low Vision Intervention Trial (LOVIT): design and methodology. Clin Trials. 2007;4(6):650-60. doi: 10.1177/1740774507085274. PMID 18042574